CLINICAL TRIAL: NCT00631007
Title: A Randomized, Double-Blind, Placebo-Controlled, 24-Week Study to Evaluate the Efficacy and Safety of INT131 Besylate Compared to Pioglitazone in Subjects With Type 2 Diabetes
Brief Title: A Placebo Controlled Safety and Efficacy Study of INT131 Besylate in Type 2 Diabetes, With an Active Comparator
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: InteKrin Therapeutics, Inc. (Industry)
Responsible Party: Chief Executive Officer, InteKrin Therapeutics Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INT131-007
Record Dates: First submitted 2008-02-27; First posted 2008-03-07 (Estimated); Results first posted 2010-09-13 (Estimated); Last update posted 2010-09-13 (Estimated); Status verified 2010-08

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 diabetes; diabetes; diabetes mellitus; diabetes mellitus, type 2; non-TZD; thiazolidinedione; selective peroxisome proliferator-activated receptor gamma modulator; SPPARM; peroxisome proliferator-activated receptor gamma; PPAR gamma; insulin sensitizer; glucose control; endocrinopathy; hypoglycemic agent; sulfonylurea; metformin; pioglitazone; nutritional and metabolic diseases
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Endocrine System Diseases; Nutritional and Metabolic Diseases | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- INT131 besylate 0.5 mg (Experimental): INT131 besylate 0.5 mg once-daily administration and matching placebo to pioglitazone HCl.
  Interventions: Drug: INT131 besylate
- INT131 besylate 1 mg (Experimental): INT131 besylate 1 mg once-daily administration and matching placebo to pioglitazone HCl
  Interventions: Drug: INT131 besylate
- INT131 besylate 2 mg (Experimental): INT131 besylate 2 mg administered once-daily and matching placebo to pioglitazone HCl
  Interventions: Drug: INT131 besylate
- INT131 besylate 3 mg (Experimental): INT131 besylate 3 mg administered once-daily and matching placebo to pioglitazone HCl
  Interventions: Drug: INT131 besylate
- pioglitazone HCl 45 mg (Active Comparator): pioglitazone HCl 45 mg administered once-daily and matching placebo to INT131 besylate
  Interventions: Drug: Pioglitazone HCl
- placebo (Placebo Comparator): placebo administered once-daily, matching placebo to INT131 besylate and matching placebo to pioglitazone HCl
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: INT131 besylate — Once-daily, oral
  Arms: INT131 besylate 0.5 mg; INT131 besylate 1 mg; INT131 besylate 2 mg; INT131 besylate 3 mg
Drug: Pioglitazone HCl — Once-daily, oral
  Other Names: Actos
  Arms: pioglitazone HCl 45 mg
Drug: Placebo — Once-daily, oral
  Arms: placebo

SUMMARY:
This is a 24 week study comparing the efficacy of four dose levels of INT131 besylate with pioglitazone HCl in patients with type 2 diabetes. Eligible patients will be men and women (of non-childbearing potential or using dual barrier methods of contraception) between 30 and 75 years of age who are minimally responsive to treatment with sulfonylurea monotherapy or sulfonylurea plus metformin combination therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Type 2 diabetes and on either sulfonylurea monotherapy or sulfonylurea plus metformin combination therapy for at least 3 months at stable dose
* Males and Females (of non-childbearing potential or who are using dual barrier methods of contraception) between 30 and 75 years of age
* HbA1c must be ≥7.5% and ≤10% at screening
* Fasting Plasma Glucose must be <240 mg/dL at screening

Exclusion Criteria:

* History of type 1 diabetes
* History of diabetic ketoacidosis
* NYHA Class III or IV cardiac status or hospitalization for congestive heart failure within 6 weeks prior to Visit 1
* Treatment with any non-peroxisome proliferator-activated receptor (non-PPAR) antidiabetic agent, investigational or approved, other than metformin or permitted sulfonylureas within 3 months prior to screening
* Treatment with rosiglitazone, pioglitazone, or any PPAR investigational antidiabetic agent within 6 month prior to screening
* Body mass index >45 kg/m2
* Fasting triglycerides >500 mg/dL
* Uncontrolled hypertension (sitting systolic blood pressure >160 mmHg and/or sitting diastolic blood pressure >100 mmHg
* Presence of diabetic complications, which in the opinion of the investigator, would complicate the subject's participation in the study (i.e., require initiation of new medication)

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 367 (Actual)
Dates: Start 2008-02; Primary Completion 2009-08 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Orloff, MD, Study Director — Medpace, Inc.
Locations (65):
- United States (58):
  - Northern California Research, Carmichael, California
  - National Research Institute, Los Angeles, California
  - VA San Diego Healthcare System, San Diego, California
  - Apex Research Institute, Santa Ana, California
  - Internal Medicine of the Rockies, Colorado Springs, Colorado
  - Creekside Endocrine Associates, PC, Denver, Colorado
  - Clinical Research Consulting, LLC, Milford, Connecticut
  - MedStar Research Institute, Washington D.C., District of Columbia
  - Clinical Research of South Florida, Coral Gables, Florida
  - The Center for Diabetes and Endocrine Care, Hollywood, Florida
  - Baptist Diabetes Associates, PA, Miami, Florida
  - International Research Associates, LLC, Miami, Florida
  - Elite Research Institute, Miami, Florida
  - Suncoast Clinical Research, Inc., New Port Richey, Florida
  - Suncoast Clinical Research, Inc., Palm Harbor, Florida
  - Meridien Research, Tampa, Florida
  - Clinical Research of Central Florida, Winter Haven, Florida
  - Executive Health and Research Associates, Inc., Atlanta, Georgia
  - Endocrine Research Solutions, Inc., Roswell, Georgia
  - Cedar-Crosse Research Center, Chicago, Illinois
  - ICCT Reseach International, Chicago, Illinois
  - American Health Network, Indianapolis, Indiana
  - L-Marc Research Center, Louisville, Kentucky
  - New Orleans Center for Clinical Research, New Orleans, Louisiana
  - Stephen R. Smith, MD, Baltimore, Maryland
  - Olive Branch Family Medical Center, Olive Branch, Mississippi
  - Diabetes and Endocrinology Specialists, Inc., Chesterfield, Missouri
  - Saint Luke's Lipid and Diabetes Reseach Center, Kansas City, Missouri
  - Bozeman Deaconess Internal Medicine Associates, Bozeman, Montana
  - Comprehensive Clinical Research, Berlin, New Jersey
  - Kaleida Health Diabetes Center, Buffalo, New York
  - UNC Diabetes Care Center/Highgate Specialty Center, Durham, North Carolina
  - Fairbrook Medical Clinic, Hickory, North Carolina
  - Diabetes & Endrocrinology Consultants, Morehead City, North Carolina
  - The Lindner Clinical Trial Center, Cincinnati, Ohio
  - IVA Research, Cincinnati, Ohio
  - Rapid Medical Research, Inc, Cleveland, Ohio
  - Opitmed Research, LTD, Columbus, Ohio
  - ResEvo LLC, Cuyahoga Falls, Ohio
  - Delaware Smith Clinic, Delaware, Ohio
  - Prestige Clinical Research, Franklin, Ohio
  - Wells Institute for Health Awareness, Kettering, Ohio
  - Frederick C Smith Clinic, Marion, Ohio
  - Your Diabetes Endocrine Nutrition Group, LLC, Mentor, Ohio
  - Clinical Research Source, Inc, Perrysburg, Ohio
  - Tri-State Medical Group, Inc., Beaver, Pennsylvania
  - Lycoming Internal Medicine, Inc., Jersey Shore, Pennsylvania
  - New England Center for Clinical Research, Cranston, Rhode Island
  - Hartwell Research Group, Anderson, South Carolina
  - Medical Research South, Charleston, South Carolina
  - Palmetto Clinical Trial Services, LLC, Simpsonville, South Carolina
  - Dallas Diabetes and Endocrine Research Center, Dallas, Texas
  - Research Institute of Dallas, Dallas, Texas
  - Baylor University Endocrine Center, Dallas, Texas
  - Diabetes Center of the Southwest, Midland, Texas
  - Quality Research, Inc., San Antonio, Texas
  - DGD Research, San Antonio, Texas
  - Salem VA Medical Center R&D Office, Salem, Virginia
- Mexico (7):
  - Nucleo Medico Vallarta, Guadalajara, Jalisco
  - Comite Mexicano para la Prevencion de la Osteoporosis A.C., Mexico City, Mexico DF
  - Centro Especializado en Diabetes y Obisidad (EDOPEC), Mexico City, Mexico DF
  - Instituto Nacional de Nutricion Salvador Zubiran (INNSZ), Mexico City, Mexico DF
  - Instituto Mexicano de Investigacion Clinica, Mexico City, Mexico DF
  - Unidad Metabolica y Cardiovascular SC, Cuernavaca, Morelos
  - Hospital Santa Engracia, Monterrey, Nuevo León

REFERENCES:
- [Derived] DePaoli AM, Higgins LS, Henry RR, Mantzoros C, Dunn FL; INT131-007 Study Group. Can a selective PPARgamma modulator improve glycemic control in patients with type 2 diabetes with fewer side effects compared with pioglitazone? Diabetes Care. 2014 Jul;37(7):1918-23. doi: 10.2337/dc13-2480. Epub 2014 Apr 10. PMID 24722496

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients 30 - 75 years of age with type 2 diabetes mellitus with inadequate glycemic control (HbA1c ≥7.5% and ≤ 10% and a Fasting Plasma Glucose <240 mg/dL) at screening on sulfonylurea monotherapy or sulfonylurea plus metformin were eligible to enter the study.
Groups:
- INT131 Besylate 0.5 mg: INT131 besylate 0.5 mg once-daily administration and matching placebo to pioglitazone.
- INT131 Besylate 1 mg: INT131 besylate 1 mg once-daily administration and matching placebo to pioglitazone
- INT131 Besylate 2 mg: INT131 besylate 2 mg administered once-daily and matching placebo to pioglitazone
- INT131 Besylate 3 mg: INT131 besylate 3 mg administered once-daily and matching placebo to pioglitazone
- Placebo: placebo administered once-daily
Period: Overall Study
Arm/Group | INT131 Besylate 0.5 mg | INT131 Besylate 1 mg | INT131 Besylate 2 mg | INT131 Besylate 3 mg | Pioglitazone HCl 45 mg | Placebo
Started | 60 | 61 | 63 | 62 | 60 | 61
Completed | 49 | 50 | 53 | 53 | 48 | 46
Not Completed | 11 | 11 | 10 | 9 | 12 | 15
Not completed — Adverse Event | 0 | 2 | 0 | 2 | 3 | 2
Not completed — Lost to Follow-up | 2 | 1 | 2 | 4 | 5 | 3
Not completed — Physician Decision | 1 | 0 | 1 | 0 | 0 | 2
Not completed — Persistent Hyperglycemia | 2 | 2 | 5 | 1 | 2 | 5
Not completed — Withdrawal by Subject | 4 | 5 | 2 | 2 | 1 | 3
Not completed — Other | 2 | 1 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | INT131 Besylate 0.5 mg | INT131 Besylate 1 mg | INT131 Besylate 2 mg | INT131 Besylate 3 mg | Pioglitazone HCl 45 mg | Placebo | Total
Number analyzed (Participants) | 60 | 61 | 63 | 61 | 60 | 61 | 366
Age Continuous [Mean (Standard Deviation); unit: years] | 54.9 (8.48) | 58.0 (9.18) | 56.1 (7.98) | 54.8 (9.76) | 55.8 (10.40) | 55.3 (10.93) | 55.8 (9.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 29 | 32 | 25 | 32 | 28 | 170
  Male | 36 | 32 | 31 | 36 | 28 | 33 | 196
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 29 | 31 | 29 | 32 | 28 | 31 | 180
  Not Hispanic or Latino | 31 | 30 | 34 | 29 | 32 | 30 | 186
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6 | 7 | 6 | 5 | 5 | 7 | 36
  Asian | 0 | 0 | 2 | 1 | 1 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 1 | 2 | 4
  Black or African American | 7 | 4 | 10 | 6 | 9 | 6 | 42
  White | 46 | 50 | 45 | 49 | 44 | 46 | 280
Region of Enrollment [Number; unit: participants]
  United States | 51 | 50 | 52 | 52 | 51 | 49 | 305
  Mexico | 9 | 11 | 11 | 9 | 9 | 12 | 61
Hemoglobin A1c [Mean (Standard Deviation); unit: Percent] | 8.3 (0.76) | 8.3 (0.71) | 8.5 (0.69) | 8.3 (0.65) | 8.2 (0.67) | 8.4 (0.80) | 8.3 (0.72)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1c (HBA1c) at Week 24 With Last Observation Carried Forward
Description: HbA1c is measured as percent. Thus this change from baseline reflects the week 24 HbA1c percent minus the Week 0 HbA1c percent
Time Frame: Weeks 0-24
Population: Randomized subjects who took at least 1 dose of double blind treatment. To be included in analysis of change from baseline to week 24 with last observation carried forward, subjects must have had baseline measurement and at least 1 post baseline measurement.
Measure: Mean (Standard Deviation); unit: Percernt
Arm/Group | INT131 Besylate 0.5 mg | INT131 Besylate 1 mg | INT131 Besylate 2 mg | INT131 Besylate 3 mg | Pioglitazone HCl 45 mg | Placebo
Number analyzed (Participants) | 60 | 59 | 61 | 60 | 58 | 58
Percernt | -0.3 (0.86) | -0.6 (0.72) | -0.9 (0.97) | -1.0 (0.80) | -0.9 (0.94) | -0.1 (0.87)

2. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 24 With Last Observation Carried Forward.
Description: The change from baseline reflects the Week 24 FPG minus the Week 0 FPG with last observation carried forward.
Time Frame: Weeks 0-24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | INT131 Besylate 0.5 mg | INT131 Besylate 1 mg | INT131 Besylate 2 mg | INT131 Besylate 3 mg | Pioglitazone HCl 45 mg | Placebo
Number analyzed (Participants) | 60 | 59 | 63 | 61 | 60 | 58
mg/dL | -0.3 (58.73) | -14.6 (48.53) | -28.9 (44.20) | -26.9 (37.23) | -33.2 (37.17) | 4.6 (41.71)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from randomization to week 26.
Arm/Group | INT131 Besylate 0.5 mg | INT131 Besylate 1 mg | INT131 Besylate 2 mg | INT131 Besylate 3 mg | Pioglitazone HCl 45 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 1/60 | 1/61 | 2/63 | 0/61 | 4/60 | 4/61
Other Adverse Events (participants affected / at risk) | 15/60 | 37/61 | 37/63 | 35/61 | 34/60 | 24/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | INT131 Besylate 0.5 mg (N=60) | INT131 Besylate 1 mg (N=61) | INT131 Besylate 2 mg (N=63) | INT131 Besylate 3 mg (N=61) | Pioglitazone HCl 45 mg (N=60) | Placebo (N=61)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-Cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pharyngeal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Spermatocele (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | INT131 Besylate 0.5 mg (N=60) | INT131 Besylate 1 mg (N=61) | INT131 Besylate 2 mg (N=63) | INT131 Besylate 3 mg (N=61) | Pioglitazone HCl 45 mg (N=60) | Placebo (N=61)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 4 | 3 | 0 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 4 | 2 | 1 | 0 | 3 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 3 | 7 | 5 | 7 | 0
Influenza (Infections and infestations) | 2 | 5 | 5 | 1 | 0 | 2
Oedema peripheral (General disorders) | 3 | 8 | 8 | 8 | 6 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 2 | 3 | 3 | 2 | 4
Urinary tract infection (Infections and infestations) | 2 | 8 | 3 | 3 | 4 | 5
Weight gain (Investigations) | 0 | 2 | 1 | 4 | 6 | 0
diarrhoea (Gastrointestinal disorders) | 1 | 2 | 2 | 3 | 3 | 4
headache (Nervous system disorders) | 0 | 5 | 3 | 5 | 3 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator and Institution shall only be permitted to publish or present the results of that portion of the Study conducted at Institution with Sponsor's prior written consent, which consent may be withheld at Sponsor's sole discretion.